CLINICAL TRIAL: NCT04719858
Title: Testing the Effectiveness of the mHealth Intervention #LIFEGOALS Targeting Health Behaviors in Early Adolescents for Promoting Mental Well-being: a Group-Randomized Controlled Trial
Brief Title: Effect of #LIFEGOALS on Adolescents' Mental Health
Acronym: MOV-E-STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Agentschap Zorg en Gezondheid, Belgium (Unknown); Vlaams Instituut Gezond Leven VZW (Unknown); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOV-E-STAR
Record Dates: First submitted 2020-12-22; First posted 2021-01-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Well-being; Life Style, Healthy; Resilience; Depressive Symptoms
Keywords: mHealth; mental well-being; adolescent; digital behavior change intervention; healthy lifestyle
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Group-Randomized Control Trial with Intervention and Control group. Randomization will occur at group level (school) to avoid spillover effects between the two conditions.
Masking Description: Participants in the intervention condition will be explained that the aim of #LIFEGOALS is to help them adopt a healthy lifestyle. The link between a healthy lifestyle and mental health may come clear when using the #LIFEGOALS app, but this will not be explained to the participants at the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group that will install the #LIFEGOALS app.
  Interventions: Behavioral: #LIFEGOALS
- Control (No Intervention): Control group that will not receive any intervention.

INTERVENTIONS:
Behavioral: #LIFEGOALS — Digital health behaviour change intervention including:
  1. self-regulation component with Fitbit: goal setting, monitoring, feedback;
  2. narrative component: every week participants receive a new episode (2-5 minutes) of a youth series modeling the target behaviours;
  3. chatbot component: automated virtual coach that will send encouraging messages and give an automated answer to user questions.
  Participants install the #LIFEGOALS app on their own mobile phone and are asked to use the app during 12 consecutive weeks. Three times per week a notification will be sent to encourage engagement with the intervention.
  Other Names: MOV-E-STAR intervention
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the effectiveness of the #LIFEGOALS intervention for promoting mental health in early adolescents.

DETAILED DESCRIPTION:
The aim of the MOV-E-STAR project is to promote mental health in early adolescents (12-15 years) by motivating them to adopt a healthy lifestyle. Adolescents can protect their mental health by increasing physical activity, reducing sitting time, getting sufficient sleep, and taking a daily breakfast. Targeting these healthy lifestyle behaviours in young adolescents is an empowering, low-threshold approach that can create large public health effects. The MOV-E-STAR project aims to meet the need for an intervention targeting these behaviors in the adolescent population. Therefore, the mobile intervention '#LIFEGOALS' was developed in collaboration with stakeholders and users. The theory-based intervention consists of an application that includes (a) a self-regulation component for goal setting, self-monitoring and feedback, (b) a narrative in the form of short episodes from a youth daily drama for modelling, attitude change and increased engagement, and (c) an automated chat-function for social support and sustained engagement with the intervention.

The current study will test the intervention in a group-randomized controlled trial for its effects on mental well-being. Participants in the intervention group will have the #LIFEGOALS intervention installed on their phone and will be asked to use the intervention for 12 consecutive weeks. Participants in the control group will not receive an intervention but will only participate in the measurements. Outcomes will be assessed at baseline, intermittent (7 weeks after baseline) and post (13 weeks after baseline). Measures will include smart wearables and surveys.

ELIGIBILITY:
Inclusion Criteria:

* General adolescent population in first, second and third year of Belgian secondary education
* Attending regular secondary education in a school in Flanders, Belgium, at time of data collection
* Good understanding of Dutch

Exclusion Criteria:

* Attending special needs education schools;
* Attending education for non-Dutch speakers.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Global Well-being from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  An overall measure of well-being and health-related quality of life will be assessed with the KIDSCREEN-10 (Erhart et al. 2009). This is a valid unidimensional global health-related quality of life index (Ravens-Sieberer et al. 2010). The KIDSCREEN-10 consists of 10 items exploring the level of the adolescent's physical activity, energy and fitness, depressive moods and stressful feelings, opportunities to structure and enjoy social and leisure time and participation in social activities, quality of interaction with parent and feelings toward parents, nature of the relation with other adolescents, and cognitive capacity and satisfaction with school performance. Items are scored on a 5-point Likert scale. Sum scores range between 10 and 50, and a higher sum score indicates better health-related quality of life. This measure of global well-being is the primary outcome measure of this study.

SECONDARY OUTCOMES:
Change in Global Well-being from Baseline to 7-week Intermittent Measurement | Baseline (Week 0) and Intermittent Measurement (Week 7)
  An overall measure of well-being and health-related quality of life will be assessed with the KIDSCREEN-10 (Erhart et al. 2009), consisting of 10 items scored on a 5-point Likert scale. The scale explores the level of the adolescent's physical activity, energy and fitness, depressive moods and stressful feelings, opportunities to structure and enjoy social and leisure time and participation in social activities, quality of interaction with parent and feelings toward parents, nature of the relation with other adolescents, and cognitive capacity and satisfaction with school performance. Sum scores range between 10 and 50, and a higher score indicates better health-related quality of life.
Change in Physical Activity (PA) from Baseline to Post-measurement | One week continuous measurement at Baseline (Week 0) and Post-measurement (Week 14)
  Average time of physical activity (PA) level (light, moderate or vigorous PA) per weekday/weekend, in minutes.
  Minutes of light, moderate and vigorous PA per day are objectively measured via Axivity trackers (accelerometers) worn at the wrist. Change in the average of light, moderate and vigorous PA from pre to post is examined for weekdays and weekend. Higher values represent more PA.
Change in Sedentary Behaviour (SB) from Baseline to Post-measurement | One week continuous measurement at Baseline (Week 0) and Post-measurement (Week 14)
  Average time seated per weekday/weekend, in minutes. Minutes of SB per day are objectively measured via Axivity trackers (accelerometers) worn at the wrist. Change in the average sedentary time from pre to post is examined for weekdays and weekend. Higher values represent more SB.
Change in Sleep Duration from Baseline to Post-measurement | One week continuous measurement at Baseline (Week 0) and Post-measurement (Week 14)
  Average time asleep per night, in hours. Sleep duration per night is objectively measured via Axivity trackers (accelerometers) worn at the wrist. Change in the average of sleep duration from pre to post is examined for nights preceding a weekday and weekend. Higher values represent more sleep.
Change in Sleep Quality from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  Sleep Quality: Average sleep quality over the past week Self-reported sleep quality will be measured in the online questionnaire via four items assessing subjective experience of sleep quality, sleep latency, sleep interruption, and daytime sleepiness. The items are based on items from 2017/18 survey of the Health Behavior in School-Aged Children (HBSC) study (Inchley, Currie, Cosma, & Samdal, 2018) and from the Adolescent Sleep Wake Scale (ASWS; Essner et al., 2015), and are scored on a 5 point Likert scale (totally disagree - totally agree). A sum-score will be calculated (ranging from 4 to 20) with higher scores indicating better perceived sleep quality.
Change in Frequency of Taking Breakfast (BF) from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  Frequency of taking breakfast, in events per week. This is assessed via 2 items from the HBSC 2017/18 study protocol (Inchley et al. 2018): one for weekdays and one for the weekend. A sum score (ranging from 0 to 7) will indicate the average days of breakfast intake per week for the last month.
Change in Psychological Well-being from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  The subscale Psychological Well-being of the KIDSCREEN-52 will assess positive emotions and satisfaction with life. This subscale consists of 6 items scored on a 5-point Likert scale. A higher sum score (ranging from 6 to 30) indicates more happiness and more positive and satisfying views of life.
Change in Moods and Emotions from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  The subscale Moods & Emotions from the KIDSCREEN-52 will assess the extent to which the adolescent experiences depressive moods and emotions and stressful feelings. This subscale consists of 7 items scored on a 5-point Likert scale. A higher sum score (ranging from 7 to 35) indicates a more positive mood and feelings.
Change in Self-Perception from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  The subscale Self-Perception from the KIDSCREEN-52 will be used to assess the perception of oneself as well as one's appearance (body image). This subscale consists of 5 items scored on a 5-point Likert scale. A higher sum score (ranging from 5 to 25) indicates greater self-confidence and self-satisfaction, and a more positive body image.
Change in Social Support and Peers from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  The subscale Social support & Peers from the KIDSCREEN-27 will be used to assess the quality of interaction with friends and peers, as well as the perceived support. This subscale consists of 4 items scored on a 5-point Likert scale. A higher sum score (ranging from 4 to 20) indicate feeling more accepted and supported.
Change in Resilience from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  Resilience will be measured by the Brief Resilience Scale (BRS) (Smith, Dalen, Wiggins, Tooley, Christopher, & Bernard, 2008). The BRS consists of 6 items scored on a 5-point Likert scale, assessing the capacity to bounce back after hard times. A higher sum score (ranging from 6 to 30) indicates greater resilience. We added a timeframe and adapted the wording of the Dutch version of the BRS (Soer et al., 2018) to make the items adequate for young adolescents. This was discussed in team, and the adapted questionnaire was tested on comprehensibility with 4 adolescents. The Dutch version of the BRS has shown sufficient reliability (α = .78) and construct validity in healthy workers (Soer et al., 2018).
Change in Depressive Symptoms from Baseline to Post-measurement | Baseline (Week 0) and Post-measurement (Week 14)
  The Custom Short Form of the Dutch version of the PROMIS Pediatric Bank v2.0 Depressive Symptoms v2.0 (PROMIS-PedDepSx; Irwin et al., 2010) will be used to assess depressive symptoms. This scale consists of 4 items scaled on a 5-point Likert scale. A higher sum score (ranging from 4 to 20) indicates more symptoms of depression. The PROMIS-PedDepSx showed good psychometric properties (Kaat et al., 2019).
Perceived Change from Baseline to Post-measurement | Post-measurement (Week 14)
  The participants' impression of change in physical activity, sedentary time, sleep time, sleep quality and breakfast will be assessed in the online questionnaires using a one-item question for each behavior: To what extent do you do this [behavior] more or less since the start of the study? Answer options range from 1 (much less) to 5 (much more).
Perceived Change from Baseline to Intermittent measurement | Intermittent measurement (Week 7)
  The participants' impression of change in physical activity, sedentary time, sleep time, sleep quality and breakfast will be assessed in the online questionnaires using a one-item question for each behavior: To what extent do you do this [behavior] more or less since the start of the study? Answer options range from 1 (much less) to 5 (much more).
Experiential Engagement with the narrative component | Only in intervention group: 1 week after installation (Week 2), Intermittent measurement (Week 7), and Post-measurement (Week 14)
  Experiential Engagement with the narrative component of the #LIFEGOALS app refers to the user's experience when watching the episodes of the narrative.
  Self-report items are based on the 'Digital Behavior Change Intervention (DBCI) engagement scale' (Perski et al., 2019). In consultation with author O. Perski, the items were adapted and limited to 3 items assessing interest, attention and affect. Items are scaled on a 5-point Likert scale. A higher sum score (ranging from 3 to 15) indicates stronger experiential engagement with the narrative.
Experiential Engagement with the remaining of the app | Only in intervention group: 1 week after installation (Week 2), Intermittent measurement (Week 7), and Post-measurement (Week 14)
  Experiential Engagement with the remaining of the #LIFEGOALS app refers to the user's experience when using the app, not considering the narrative.
  Self-report items are based on the 'Digital Behavior Change Intervention (DBCI) engagement scale' (Perski et al., 2019). In consultation with author O. Perski, the items were adapted and limited to 4 items assessing interest, attention, affect and usability. Items are scaled on a 5-point Likert scale. A higher sum score (ranging from 4 to 20) indicates stronger experiential engagement with the rest of the app.
Behavioral Engagement | Only in intervention group: Continuous assessment throughout the 12 weeks of intervention.
  Behavioral Engagement with the #LIFEGOALS app refers to the actual usage of the app.
  It is assessed by logging user's activity in the app. Out of the system log data, the duration of usage will be extracted. Behavioral engagement will be reported as the average minutes of usage per week.

OTHER OUTCOMES:
Age | Baseline (Week 0)
  Calculated on birthday
Gender | Baseline (Week 0)
  'girl', 'boy' or 'other'
Type of education | Baseline (Week 0)
  general, technical or vocational
Grade | Baseline (Week 0)
  1st, 2nd or 3th grade of highschool
Socio-economic status | Baseline (Week 0)
  Family Affluence measured with the Family Affluence Scale (FAS, Health-Behavior in School-Aged Children study 2017-2018) questionnaire consisting of 6 items. These items are combined to produce a composite score ranging from 0 (low affluence) to 9 (high affluence).
  Highest Diploma of Father; Highest Diploma of Mother; Language spoken at home; Job of Father; Job of Mother; Subjective Experience of Financial Situation;
Change in Attitude from Baseline to Intermittent and Post measurement | Baseline (Week 0), Intermittent measurement (Week 7), and Post-measurement (Week 14)
  Attitude regarding PA, SB, SL and BF is assessed in the online surveys using 3 items for each of the four behaviors. Items are scaled on a 5-point Likert scale. Items were pretested in a pilot study. Higher sum scores indicate higher self-reported attitude.
Change in Self-efficacy from Baseline to Intermittent and Post measurement | Baseline (Week 0), Intermittent measurement (Week 7), and Post-measurement (Week 14)
  Self-efficacy regarding PA, SB, SL and BF is assessed in the online surveys using 3 items for each of the four behaviors. Items are scaled on a 5-point Likert scale. Items were pretested in a pilot study. Higher sum scores indicate higher self-reported self-efficacy.
Change in Intention from Baseline to Intermittent and Post measurement | Baseline (Week 0), Intermittent measurement (Week 7), and Post-measurement (Week 14)
  Participants' intention for PA, reduced SB, sufficient SL and daily BF is assessed in the online surveys using 1 item for each of the four behaviors. Items are scaled on a 5-point Likert scale. Items were pretested in a pilot study. Higher scores indicate higher self-reported intention.

CONTACTS AND LOCATIONS:
Overall Officials: Greet Cardon, Prof, Principal Investigator — University Ghent; Geert Crombez, Prof, Principal Investigator — University Ghent; Ann DeSmet, PhD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
During the study, only the researchers that are involved in the study will have access to the full data of the participants, only for research purposes.
  After the study, anonymized data will be shared with other researchers within our research group, and will be made available to other researchers upon request.
  After publication of the study results, the data will be made accessible on the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol will be registered on OSF in January 2021. The collected data will be shared upon request for 5 years after the study has finished (June 2020).
  Data and statistical analyses that underlie results in a publication will be placed on OSF upon acceptation of the manuscript.
Access Criteria: Supporting information underlying results in a publication will be made publically available (OSF). Other supporting information will be made available to other researchers upon request.

REFERENCES:
- [Derived] Peuters C, Maenhout L, Cardon G, De Paepe A, DeSmet A, Lauwerier E, Leta K, Crombez G. A mobile healthy lifestyle intervention to promote mental health in adolescence: a mixed-methods evaluation. BMC Public Health. 2024 Jan 2;24(1):44. doi: 10.1186/s12889-023-17260-9. PMID 38166797
- [Derived] Maenhout L, Peuters C, Cardon G, Crombez G, DeSmet A, Compernolle S. Nonusage Attrition of Adolescents in an mHealth Promotion Intervention and the Role of Socioeconomic Status: Secondary Analysis of a 2-Arm Cluster-Controlled Trial. JMIR Mhealth Uhealth. 2022 May 10;10(5):e36404. doi: 10.2196/36404. PMID 35536640